CLINICAL TRIAL: NCT06126289
Title: Cerebrospinal Fluid Single-cell Sequencing and Proteomics Analysis of the Chronic Postsurgical Pain in Patients Following Open Reduction Internal Fixation of Lower Limb Fractures
Brief Title: CSF Single-cell Sequencing and Proteomics of Chronic Postsurgical Pain in Patients With Lower Limb Fractures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XZXY-LK-20230530-084
Record Dates: First submitted 2023-10-31; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-06

CONDITIONS: Chronic Postsurgical Pain
Keywords: Chronic Postsurgical pain; Single-cell sequencing; Cerebrospinal Fluid
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients undergoing hardware removal following open reduction internal fixation of lower limb fractures under spinal anesthesia will be enrolled in the study. The anesthesiologist retained cerebrospinal fluid during a subarachnoid puncture.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pain-free control subjects: According to the 11th Revision of International Classification of Diseases (ICD-11) of International Association for the Study of Pain(IASP) in 2019, diagnose whether patients have CPSP . Patients with no postoperative chronic pain after open reduction and internal fixation of lower limb fractures.
- Patients with chronic postsurgical pain: According to the 11th Revision of International Classification of Diseases (ICD-11) of International Association for the Study of Pain(IASP) in 2019, diagnose whether patients have CPSP . Patients with postsurgical chronic pain after open reduction and internal fixation of lower limb fractures.

SUMMARY:
The purpose of this study is to assess the proteomics and transcriptomic differences between pain-free control subjects and patients with chronic postoperative pain through single-cell sequencing technology.

DETAILED DESCRIPTION:
Chronic pain,one of the most frequent causes for patients to seek medical care,is a recognized health problem.Chronic postsurgical pain (CPSP), commonly defined as pain that develops after a surgical procedure and persists at least 3 months, constitutes a widely underdiagnosed and often poorly treated medical problem affecting 10-50% of all postsurgical patients. According to the reports,in the United States alone,1.9 million persons abused or were dependent on prescription opioid analgesics for chronic pain in 2013,contributing to one of the worst public health crises the developed world has recently faced.Here,open reduction and internal fixation of lower limb fractures ,what we focus, is a common surgical procedure in orthopedics and microscopic hand and foot surgery.The removal of the intramedullary nail can relieve anterior knee pain, but in a substantial number of patients, pain persists after nail removal.The most painful daily activities are kneeling and squatting.Therefore, it is increasingly important and urgent to solve the postoperative chronic pain of patients with lower extremity fractures surgery.

The underlying biology of chronic postoperative pain and genetic heritability is complex and not yet fully understood . A common feature of CPSP is that the painful sensations change from the familiar acute postoperative pain to a complex pain syndrome with nociplastic characteristics,neuropathic characteristics, or both. Preclinical studies have revealed that neuroinflammation is one of pathological hallmarks of CPSP. The transition from acute to chronic pain starts early within the first 2 weeks after nociception by peripheral and central inflammatory processes and activation of spinal glial cells.Repetitive nociception resulting from prolonged inflammatory and neuropathic responses to noxious stimuli causes a cascade of biochemical and structural changes to various pain pathways resulting in sensitization of the peripheral and CNS. Cytokines and neurotrophic factors have been identified as pivotal mediators involved in neuroimmune activation pathways and cascades in various preclinical chronic pain models.

The brain is surrounded by the meninges, a membranous covering that contains the cerebrospinal fluid (CSF).Its circulatory system transmits peripheral stimulation to the cerebrum, and central signal is transmitted to the dorsal root ganglion. CSF ,as a bridge between peripheral and central, contains a tightly regulated immune system and metabolitites and reflects the inflammatory processes and activation of spinal glial cells. However, knowledge is lacking about how CSF contains are altered with pain.We thus hypothesized that comparing the CSF protemics and immune transcriptomes associated with pain-free control subjects and patients with chronic postoperative pain would provide insights into the pathophysiology of CPSP. Here,a single-cell transcriptomic resource exploring the cerebrospinal fluid immune system and proteomics of patients with postoperative chronic pain will uncover the key molecules and pathways of CPSP.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status 1 to 3 (males and females)
2. Undergone open reduction and internal fixation of the lower limbs and plan to take out the internal fixation under spinal anesthesia

Exclusion Criteria:

1. Absence of written consent
2. Contraindication to regional anaesthesia
3. Known dementia at time of operation
4. History or opioid abuse
5. Unexpected conversion of general anesthesia or surgery is not carried out

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had undergone open reduction and internal fixation of the lower limbs and planned to take out the internal fixation were interviewed before surgery to collect the basic data ( gender, age, BMI, etc. ) and previous surgical information. Selecting the patients with the chronic postoperative pain，for one-to-one case matching.All patients and control subjects were without any analgesic medicatio during the 24hours before the investigation,and were not using any daily mediciation.Routine blood and urine assessments were within the normal range.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-12-25 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Significantly different proteomics and transcriptomes between Chronic Postsurgical Pain and pain-free subjects | Up to 3 months after fixation
  Differences in the proteins in the fluid around the lumbar, between Chronic Postsurgical Pain and Pain-free subjects.，will be quantified using Mass spectrometry，for:
  neural cell adhesion molecule L1, complement C4-A, lysozyme C, receptor-type tyrosine-protein phosphatase zeta, apolipoprotein D, alpha-1-antichymotrypsin, granulins, calcium/calmodulin-dependent protein kinase type II subunit alpha, mast/stem cell growth factor receptor Kit, prolow-density lipoprotein receptor-related protein 1 and so on.
  These proteins may identify the disease and define its mechanism.
Inflammatory cytokines in Chronic Postsurgical Pain patients | Up to 3 months after fixation surgery
  Biomarkers from CSF will be quantified using Meso Scale Discovery multiplex kit (K15210D), for:
  CRP, Eotaxin, Eotaxin-3, FGF (basic), ICAM-1, IFN-γ, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12/IL-23p40, IL-13, IL-15, IL-16, IL-17A, IP-10, MCP-1, MCP-4, MDC, MIP-1α, MIP-1β, PlGF, SAA, TARC, Tie-2, TNF-α, TNF-β, VCAM-1, VEGF-A, VEGF-C, VEGF-D, VEGFR-1/Flt-1.
  The levels of these biomarkers will be compared between the group between CPSP and pain-free subjects.

REFERENCES:
- [Background] Scholz J, Finnerup NB, Attal N, Aziz Q, Baron R, Bennett MI, Benoliel R, Cohen M, Cruccu G, Davis KD, Evers S, First M, Giamberardino MA, Hansson P, Kaasa S, Korwisi B, Kosek E, Lavand'homme P, Nicholas M, Nurmikko T, Perrot S, Raja SN, Rice ASC, Rowbotham MC, Schug S, Simpson DM, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ, Barke A, Rief W, Treede RD; Classification Committee of the Neuropathic Pain Special Interest Group (NeuPSIG). The IASP classification of chronic pain for ICD-11: chronic neuropathic pain. Pain. 2019 Jan;160(1):53-59. doi: 10.1097/j.pain.0000000000001365. PMID 30586071
- [Background] van Ransbeeck A, Budilivski A, Spahn DR, Macrea L, Giuliani F, Maurer K. Pain Assessment Discrepancies: A Cross-Sectional Study Highlights the Amount of Underrated Pain. Pain Pract. 2018 Mar;18(3):360-367. doi: 10.1111/papr.12612. Epub 2017 Sep 20. PMID 28707777
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Clay FJ, Watson WL, Newstead SV, McClure RJ. A systematic review of early prognostic factors for persisting pain following acute orthopedic trauma. Pain Res Manag. 2012 Jan-Feb;17(1):35-44. doi: 10.1155/2012/935194. PMID 22518366
- [Background] Friesgaard KD, Gromov K, Knudsen LF, Brix M, Troelsen A, Nikolajsen L. Persistent pain is common 1 year after ankle and wrist fracture surgery: a register-based questionnaire study. Br J Anaesth. 2016 May;116(5):655-61. doi: 10.1093/bja/aew069. PMID 27106969
- [Background] Leliveld MS, Van Lieshout EMM, Polinder S, Verhofstad MHJ; TRAVEL Study Investigators. Effect of Transverse Versus Longitudinal Incisions on Anterior Knee Pain After Tibial Nailing (TRAVEL): A Multicenter Randomized Trial with 1-Year Follow-up. J Bone Joint Surg Am. 2022 Dec 21;104(24):2160-2169. doi: 10.2106/JBJS.22.00389. Epub 2022 Oct 25. PMID 36367768
- [Background] Rees S, Tutton E, Achten J, Bruce J, Costa ML. Patient experience of long-term recovery after open fracture of the lower limb: a qualitative study using interviews in a community setting. BMJ Open. 2019 Oct 9;9(10):e031261. doi: 10.1136/bmjopen-2019-031261. PMID 31601595
- [Background] Fitzcharles MA, Cohen SP, Clauw DJ, Littlejohn G, Usui C, Hauser W. Nociplastic pain: towards an understanding of prevalent pain conditions. Lancet. 2021 May 29;397(10289):2098-2110. doi: 10.1016/S0140-6736(21)00392-5. PMID 34062144
- [Background] Hankerd K, McDonough KE, Wang J, Tang SJ, Chung JM, La JH. Postinjury stimulation triggers a transition to nociplastic pain in mice. Pain. 2022 Mar 1;163(3):461-473. doi: 10.1097/j.pain.0000000000002366. PMID 34285154
- [Result] Wyss-Coray T, Mucke L. Inflammation in neurodegenerative disease--a double-edged sword. Neuron. 2002 Aug 1;35(3):419-32. doi: 10.1016/s0896-6273(02)00794-8. PMID 12165466